CLINICAL TRIAL: NCT05946876
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics of XH-S003 After Single and Multiple Ascending Doses, Plus the Evaluation of Food Effects in Healthy Volunteers
Brief Title: A Phase 1 Study of XH-S003 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S-INFINITY Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-S003-101
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (XH-S003) (Experimental): Participants will receive an oral dose of XH-S003 once daily on scheduled day(s).
  Dosage: Part A : 50mg,100mg, 200mg, 25mg & 400mg Part B : 25mg, 50mg, 100mg. Part C : 200 mg
  Interventions: Drug: XH-S003 (A)
- B (Placebo) (Placebo Comparator): Participants will receive oral matching placebo once daily on scheduled day(s)
  Interventions: Other: Placebo (B)

INTERVENTIONS:
Drug: XH-S003 (A) — IP: XH-S003 IP: XH-S003 Dose: 25 mg, 100 mg Dose Formulation: Capsule Route of Administration: Oral
  Arms: A (XH-S003)
Other: Placebo (B) — Dose: 25 mg, 100 mg Dose Formulation: Capsule Route of Administration: Oral
  Arms: B (Placebo)

SUMMARY:
This is a phase 1, randomised, first-in-human, double-blinded, placebo-controlled, SAD (Single Ascending Dose) and MAD (Multiple Ascending Dose) study to assess the PK, safety, and tolerability of XH-S003 in healthy volunteers. In addition, this study evaluates the effects of food on XH-S003 under a two-period, cross-over study setting.

DETAILED DESCRIPTION:
The study is composed of three parts. Part A (SAD portion, 5 cohorts) and Part B (MAD portion, 3 cohorts) of the study will enrol eligible participants and provide various doses of XH-S003 or placebo at a ratio of 3:1 in each cohort. Part C of the study plans to evaluate the food effect on XH-S003.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 to ≤ 55 years old.
2. BMI between ≥ 19.0 and ≤ 30.0 kg/m2 at Screening, and weight between ≥ 50 kg and ≤ 120.0kg for male, weight ≥ 45 kg and ≤ 120.0kg for female.
3. Able and willing to comply with the study procedure and the restriction specified in the protocol.
4. Provision of signed and dated written informed consent prior to any study specific procedures.
5. Female subjects of childbearing potential must have a negative serum pregnancy test result at screening and a negative pregnancy test result at baseline, and agree to use one of the acceptable methods of contraception listed below during the study (from the time of signing the informed consent until one month after the end of study [EOS] or early termination visit evaluation [ET]):

   * The subject's male partner has undergone documented vasectomy with documentation of azoospermia (male sterilization).
   * A documented placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Consistent use of the same oral contraceptives for at least 3 months before screening, injectable progesterone, subdermal implants, or the use of a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps], which present no effect on IP at the discretion of investigator).
   * Documented tubal ligation (female sterilization).
   * True abstinence: when this is in line with the preferred and usual lifestyle of the subject, including female subjects with same sex partners. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects must agree to use one of the above-mentioned contraceptive methods, if they start sexual relationships during the study.
6. Male subjects agreeing to use acceptable methods of contraception if the male subject's partner could become pregnant from the time of signing the informed consent until 3 months after EOS/ET. One of the following acceptable methods of contraception must be utilized:

   * Surgical sterilization (vasectomy with documentation of azoospermia).
   * The subject's female partner uses oral contraceptives (including combination estrogen/progesterone pills, progesterone pills), injectable progesterone, or subdermal implants, or a barrier method (condom or occlusive cap [diaphragm or cervical/vault caps]).
   * The subject's female partner uses medically prescribed topically applied transdermal contraceptive patch.
   * The subject's female partner has undergone documented tubal ligation (female sterilization).
   * The subject's female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * True abstinence: when this is in line with the preferred and usual lifestyle of the subject, including male subjects with same sex partners. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects must agree to use one of the above-mentioned contraceptive methods, if they start sexual relationships during the study.
7. Subjects do not plan to donate sperm or eggs from the time of signing the informed consent until 3 months after EOS/ET.

Exclusion Criteria:

1. Subjects with a history of allergies to similar ingredients of the study drug or any ingredient in the study drug, or vaccine component; subjects with a history of severe allergic or anaphylactic reactions at the discretion of PI. Subjects with one of the conditions (including, but not limited to):

   * Subjects with history of eczema within 3 years.
   * Subjects with asthma except for resolved childhood asthma.
   * Subjects with clinical syndromes of urticaria at screening or baseline.
2. Subjects whose abnormalities in past medical history are clinically significant or other clinical findings suggest the following clinically significant diseases at the discretion of the PI (including but not limited to gastrointestinal, renal, hepatic, neurological, hematologic, endocrine, pulmonary, psychiatric, or cardiovascular and cerebrovascular diseases, which are deemed as clinically significant by PI).
3. Abnormal liver function tests at screening, defined as alanine aminotransferase (ALT) or aspartate transaminase (AST) > 1.5x upper limit of normal (ULN), and bilirubin >1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) that are considered by the PI to be clinically significant. Repeat tests are permitted at investigator discretion.
4. Abnormal ECG findings at Screening or Day -1 (eg, repeated demonstration of a QTc interval > 450 ms [male] or > 470 ms [female] corrected by Fridericia's formula [QTcF] or Bazett's formula [QTcB]; heart rate [HR] is out of normal range 45-100 bmp; PR is out of normal range 120 -220 msec; QRS is out of normal range <120msec) that are considered by the PI or designee to be clinically significant. Repeat tests are permitted at investigator discretion.
5. Subjects with clinically significant infection (e.g., requiring hospitalization or parenteral antimicrobial therapy) within 2 months before screening or active systemic bacterial, viral, or fungal infection or fever with ear temperature > 37.7℃ within 2 weeks before screening at the discretion of the PI.
6. Known or suspected immunodeficiency, hereditary or acquired complement deficiency.
7. Clinical laboratory evidence or clinical diagnosis of human immunodeficiency virus (HIV) infection, hepatitis C virus (HCV) infection, or chronic hepatitis B virus (HBV) infection (as shown by hepatitis B surface antigen [HBsAg] positivity).
8. Subjects who had major injuries or underwent major surgery or had not recovered from surgery or had the surgery affecting the drug metabolic process and safety assessment within 6 months prior to screening, or who are scheduled to undergo surgery during the study period.
9. Donated more than 400 mL of blood within 90 days or donated plasma within 14 days before screening.
10. Subjects who received blood product transfusion within 90 days before screening.
11. Used any medications (including but not limited to prescription medication, over-the-counter medication, herb, etc. [except for contraceptive use]) within 14 days or 7 half-lives (whichever is longer) of administration of the first dose of investigational product.
12. Subjects positive for drug abuse test or with a history of drug abuse at screening. One repeat test on the same day is permitted.
13. Subjects with a history of alcohol abuse within 1 month prior to screening (average consuming 14 units or more of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 125 mL of wine) or positive for alcohol breath test (one repeat test on the same day is permitted) at screening.
14. Subjects who smoked more than 5 cigarettes every day within 1 month prior to screening or who are not willing to quit smoking during the confinement.
15. Subjects who consume food or beverage containing grapefruit/pomelo or alcohol/caffeine (e.g., coffee, chocolate, cola, tea, etc.) within 48 hours prior to confinement and during the confinement.
16. Subjects who are unable to avoid strenuous exercise during confinement.
17. Subjects who have participated in other drug clinical trials within 3 months prior to screening or plan to participate in other clinical trial from enrolment to EOS/ET.
18. Subjects who are not suitable for venous blood collection.
19. Any other conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrolment or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part A: Upto 10 days
  AEs assessed based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of participants with adverse events (AEs) | Part B: Up to 28 days
  AEs assessed based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of participants with adverse events (AEs) | Part C: Up to 7 days
  AEs assessed based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Number of participants with clinical laboratory abnormalities | Part A: Upto 10 days
Number of participants with clinical laboratory abnormalities | Part B: Up to 28 days
Number of participants with clinical laboratory abnormalities | Part C: Up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia